CLINICAL TRIAL: NCT00414765
Title: Open-label Pharmacokinetic Trial of Aldesleukin (Rh-Interleukin-2 [IL-2]) Administered Intravenously to Subjects With Metastatic Renal Cell Carcinoma or Metastatic Melanoma With Immunologic Correlative Studies
Brief Title: Aldesleukin in Participants With Metastatic Renal Cell Carcinoma or Metastatic Melanoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPRL002A2201
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Melanoma
Keywords: Metastatic Renal Cell Carcinoma; Metastatic Melanoma; Aldesleukin; IL-2
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aldesleukin (Experimental): All participants were treated with aldesleukin 600,000 international units per kilogram [IU/kg] (0.037 milligram (mg)/kg) administered as a 15-minute intravenous (IV) infusion every 8 hours for a maximum of 14 doses for the first cycle (5-day cycle). Following 9 days of rest from therapy, the cycle was repeated for up to 14 doses (i.e., a total of up to 28 doses), if tolerated.
  Interventions: Drug: Aldesleukin

INTERVENTIONS:
Drug: Aldesleukin
  Other Names: Proleukin®; PRL002

SUMMARY:
This study evaluated the pharmacokinetics of aldesleukin in participants with metastatic renal cell cancer or metastatic melanoma.

ELIGIBILITY:
Inclusion criteria:

* Performance Status Eastern Cooperative Oncology Group: 0 or 1.
* Adequate organ function.

Exclusion criteria:

* Pregnancy or lactation.
* Prior treatment with any form of IL-2.
* Organ transplant. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2010-03-28 (Actual); Study Completion 2010-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - USC/Kenneth Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 4 investigative sites in the United States from 03-September-2008 to 28-March-2010.
Pre-assignment Details: A total of 26 participants were enrolled in the study. The study consisted of two cycles of aldesleukin, each cycle consisted of a 5-day period and a 9-day rest period between cycles.
Groups:
- mRCC Group: Participants with metastatic renal cell carcinoma (mRCC) were administered aldesleukin 600,000 IU/kg (0.037 mg/kg) as a 15-minute IV infusion every 8 hours for a maximum of 14 doses for the first cycle (5-day cycle). Following 9 days of rest from therapy, the cycle was repeated for up to 14 doses (i.e., a total of up to 28 doses), if tolerated.
- Metastatic Melanoma Group: Participants with metastatic melanoma were administered aldesleukin 600,000 IU/kg (0.037 mg/kg) as a 15-minute IV infusion every 8 hours for a maximum of 14 doses for the first cycle (5-day cycle). Following 9 days of rest from therapy, the cycle was repeated for up to 14 doses (i.e., a total of up to 28 doses), if tolerated.
Period: Overall Study
Arm/Group | mRCC Group | Metastatic Melanoma Group
Started | 7 | 19
Completed Study (A participant was considered a completer when the participant did not die or have disease progression at the end of treatment.) | 7 | 18
Completed Cycle 1 (Completion of a cycle was defined as any participant who received at least seven IV infusions during the cycle.) | 7 | 19
Completed Cycle 2 (Completion of a cycle was defined as any participant who received at least seven IV infusions during the cycle.) | 4 | 16
Completed | 1 | 8
Not Completed | 6 | 11
Not completed — Adverse Event | 5 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety set consisted of all participants who received at least one dose of aldesleukin and had at least one post-baseline safety assessment.
Groups:
- mRCC Group: Participants with mRCC were administered aldesleukin 600,000 IU/kg (0.037 mg/kg) as a 15-minute IV infusion every 8 hours for a maximum of 14 doses for the first cycle (5-day cycle). Following 9 days of rest from therapy, the cycle was repeated for up to 14 doses (i.e., a total of up to 28 doses), if tolerated.
- Total: Total of all reporting groups
Arm/Group | mRCC Group | Metastatic Melanoma Group | Total
Number analyzed (Participants) | 7 | 19 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (4.68) | 51.3 (12.08) | 53.2 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in the Area Under the Concentration-Time Curve (AUC) From 0 to 8 Hours (AUC0-8) of Aldesleukin After One Cycle of Therapy
Time Frame: From Cycle 1, Day 1 to Cycle 2, Day 15
Population: The Pharmacokinetic Analysis (PK) set consisted of all participants in the safety set who completed two cycles of aldesleukin therapy and had evaluable post-baseline blood samples on Cycle 1, Day 1 and Cycle 2, Day 15. The Safety set consists of all participants who received at least one dose of aldesleukin and had at least one post-baseline safety assessment.
Measure: Mean (Standard Deviation); unit: hour times picograms per mL(h × pg/mL)
Arm/Group | mRCC Group | Metastatic Melanoma Group
Number analyzed (Participants) | 2 | 11
hour times picograms per mL(h × pg/mL)
  Participants With Presence of Anti-IL-2 antibodies (Anti-IL-2 Ab) Titer: number analyzed (Participants) | 2 | 9
  Participants With Presence of Anti-IL-2 antibodies (Anti-IL-2 Ab) Titer | 60359.9 (37406.04) | 173127.7 (223655.01)
  Participants With Absence of Anti-IL-2 Ab Titer: number analyzed (Participants) | 0 | 2
  Participants With Absence of Anti-IL-2 Ab Titer |  | -22171.6 (14798.46)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to approximately 47 days.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus 28 days post treatment.
Groups:
- mRCC: mRCC
- Metastatic Melanoma: Metastatic Melanoma
Arm/Group | mRCC | Metastatic Melanoma
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/7 | 4/19
Other Adverse Events (participants affected / at risk) | 0/7 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mRCC (N=7) | Metastatic Melanoma (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.